CLINICAL TRIAL: NCT00739440
Title: Randomized Controlled Trial to Evaluate Efficiency and Safety of the Polyvalent Antiscorpion Serum of Birmex Versus Other Commercial Serum
Brief Title: Randomized Controlled Trial to Compare Two Anti-scorpion Serums
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios de Biologicos y Reactivos de México, S.A. de C.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Birmex-01-2008
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Scorpion Sting
MeSH Terms: conditions — Scorpion Stings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Patients 15 to 60 years with scorpion sting, will receive serum antiscorpion elaborated by Birmex
  Interventions: Biological: serum antiscorpion
- II (Experimental): Patients 15 to 60 years with scorpion sting, will receive other commercial serum antiscorpion (Alacramyn)
  Interventions: Biological: serum antiscorpion

INTERVENTIONS:
Biological: serum antiscorpion — The dose may be required for the patient according to clinical manifestations and evolution
  Other Names: anti-Scorpion venom Serum

SUMMARY:
The purpose of this study is to compare the efficiency and safety of the treatment against sting scorpion, using two serums, one elaborated by Birmex versus other commercial serum

DETAILED DESCRIPTION:
We consider relevant conduct this study because the poisoning scorpion bite represents a public health problem.

This is a randomized clinical trial, which included 120 subjects of both sexes aged 15 and 60 years old and residents of the state of Guanajuato, divided into 2 groups: 60 patients received antiscorpion serum of Birmex and 60 patients receive other commercial serum.

ELIGIBILITY:
Inclusion Criteria:

* Sting scorpion
* Informed consent
* Age 15-60
* Either sex
* Resident in study area

Exclusion Criteria:

* Previous treatment with gammaglobulin
* Blood transfusion at any stage of life
* Sensitivity or intolerance to serums antiscorpion or horse products
* Pregnancy
* Some immunodeficiency

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Resolution of signs and symptoms of scorpion envenomation | after treatment (expected average of 12 hrs)

SECONDARY OUTCOMES:
Evaluate the adverse events in every treated child | inmediately after treatment and until 5 days later

CONTACTS AND LOCATIONS:
Overall Officials: Jimenez C Ma. Eugenia, PhD, Principal Investigator — Laboratorios de Biologicos y Reactivos de México, S.A. de C.V.